CLINICAL TRIAL: NCT05933213
Title: Comparing Efficacy and Safety of Mescaline Sodium Enteric-coated Tablets vs Morte-mescaline in the Treatment of Adult Lupus Nephritis: A Prospective, Multicenter,Real-world Study
Brief Title: Comparing Mescaline Sodium Enteric-coated Tablets vs Morte-mescaline in the Treatment of Adult Lupus Nephritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Beijing Medical Award Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXJL-2023-0532-0027
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; mescaline sodium enteric-coated tablets; morte-mescaline
MeSH Terms: conditions — Lupus Nephritis | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mescaline sodium enteric-coated tablets group (Experimental): Treating with glucocorticoids + mescaline sodium enteric-coated tablets
  (1) Induction period: Prednisone tablets: orally, recommended dose 0.4-0.8 mg/kg/d, with gradual dose reduction (10% per month) at the end of 3-6 months; mescaline sodium enteric-coated tablets: orally, twice a day, at 720-1440 mg/d, for 3-6 months; (2) Maintenance period: Prednisone tablets 5-7.5 mg/d, mescaline sodium enteric-coated tablets 360-540mg/d, maintenance treatment for 1 year
  Interventions: Drug: Mescaline sodium enteric-coated tablets; Drug: Glucocorticoids
- Morte-mescaline group (Active Comparator): Treating with glucocorticoids + morte-mescaline
  1. Induction period: Prednisone tablets: oral, recommended dose 0.4-0.8 mg/kg/d, with gradual dose reduction (10% per month) at the end of 3-6 months; mortifamate: oral, twice a day, dose 1-2 g/d, 3-6 months;
  2. Maintenance period: Prednisone tablets 5-7.5 mg/d, mortifamate 0.5-0.75 g/d, with maintenance treatment for 1 year.
  Interventions: Drug: Morte-mescaline; Drug: Glucocorticoids

INTERVENTIONS:
Drug: Mescaline sodium enteric-coated tablets — Induction period: orally, twice a day, at 720-1440 mg/d； Maintenance period: orally, twice a day, 360-540mg/d
  Arms: Mescaline sodium enteric-coated tablets group
Drug: Morte-mescaline — Induction period: orally, twice a day, 1-2 g/d; Maintenance period: orally, twice a day, 0.5-0.75 g/d
  Arms: Morte-mescaline group
Drug: Glucocorticoids — glucocorticoids

SUMMARY:
The goal of this prospective, multicenter,real-world study is to To evaluate the efficacy and safety of mescaline sodium enteric-coated tablets versus morte-mescaline in the treatment of adult patients with lupus nephritis under real-life medical conditions.

The main question it aims to answer are: Is the efficacy of mescaline sodium enteric-coated tablets in the treatment of adult patients with lupus nephritis not inferior to morti-mescaline？ Participants will receive induction and maintenance treatment with mescaline sodium enteric-coated tablets and morte-mescaline.Then participants will be followed up at 60, 180, 270 and 540 days of treatment to assess the efficacy and safety of mescaline sodium enteric-coated tablets compared to morte-mescaline.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-70 years; 2. Meet the 2019 SLE classification criteria established by EULAR/ACR; 3. Have any of the following clinical and laboratory abnormalities: 1) proteinuria >0.5 g/24h, or urine protein ++++ on random urinalysis, or urine protein/creatinine ratio EE >500 mg/g (50 mg/mmol); 2) cellular tubularity including erythrocyte tubularity, hemoglobin tubularity, granular tubularity, tubular tubularity, or mixed tubularity; 3) active urinary sediment (except 3) active urine sediment (except urinary tract infection, urine leukocytes >5/HPF, urine red blood cells >5/HPF), or erythrocyte tubular, or leukocyte tubular; 4. 24h urine protein quantification ≥ 1.0 g; 5. Require long-term treatment with MPA-type drugs (mescaline sodium enteric-coated tablets or morte-mescaline); 6. Singed the informed consent.

Exclusion Criteria:

* 1. Patients treated with immunosuppressive agents (e.g. CTX, MPA, CNI, etc.) within 30 days 2. Patients with co-morbid severe CNS infections 3. Neutrophil counts <1×103/µl; 4. Glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 ; 5. Glutamic aminotransferase (ALT), glutamic oxalacetic aminotransferase (AST) or total bilirubin > 1.5 x upper limit of normal (ULN); 6. Pregnant or lactating women 7. Presence of other major diseases such as tumors, HIV viral infections, systemic bacterial/fungal/viral infections; 8. Presence of contraindications to glucocorticoids and investigational drugs 9. Any condition that, in the judgment of the investigator, is unstable or may jeopardize the safety of the subject and his or her compliance with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2023-07-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total effective rate | 180 days of treatment
  (Complete remission + Partial remission) / total number of cases

SECONDARY OUTCOMES:
Overall incidence of adverse events and serious adverse reactions | 540 days of treatment
  Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: LUO HUI, Doctor, Principal Investigator — Xiangya Hospital of Central South University

IPD SHARING:
Plan to Share IPD: Undecided